CLINICAL TRIAL: NCT01991483
Title: A Multiple-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY2928057 in Hemodialysis Patients
Brief Title: A Study of LY2928057 in Hemodialysis Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15268; I5M-MC-FABC (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Results first posted 2019-02-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Renal Insufficiency, Chronic; Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY2928057 (No ESA) (Experimental): Multiple doses of LY2928057 administered intravenously (IV) either once every 2 weeks (Q2W) or once per week (QW) for 6 weeks. Participants discontinued their personal physician-prescribed erythropoiesis stimulating agent (ESA) before treatment.
  Interventions: Drug: LY2928057
- LY2928057 (Reduced ESA) (Experimental): Multiple doses of LY2928057 administered IV either Q2W or QW for 6 weeks. Participants reduced their personal physician-prescribed ESA dose before treatment.
  Interventions: Drug: LY2928057
- Placebo (No ESA) (Placebo Comparator): Multiple doses of placebo administered IV either Q2W or QW for 6 weeks. Participants discontinued their personal physician-prescribed ESA dose before treatment.
  Interventions: Drug: Placebo
- Placebo (Reduced ESA) (Placebo Comparator): Multiple doses of placebo administered IV either Q2W or QW for 6 weeks. Participants reduced their personal physician-prescribed ESA dose before treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2928057 — Administered intravenously
  Arms: LY2928057 (No ESA); LY2928057 (Reduced ESA)
Drug: Placebo — Administered intravenously
  Arms: Placebo (No ESA); Placebo (Reduced ESA)

SUMMARY:
This study will evaluate the safety of LY2928057 and how LY2928057 affects hemoglobin in hemodialysis participants. This study will involve multiple doses of LY2928057 given during a 6 week period either after a participant discontinues or reduces treatment to stimulate red blood cells. This study will last up to 26 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants having end-stage renal disease (ESRD), have received an erythropoiesis stimulating agent (ESA) at least weekly for 2 weeks prior to screening, and have been receiving adequate maintenance hemodialysis (3 times weekly) for at least 12 weeks prior to screening (that is, an approximate Kt/V greater than 1.1 (K equals dialyzer clearance of urea, t equals dialysis duration time, V equals volume of distribution of urea, which is approximately equal to the participant's total body water) based on the clinical judgment of participant's nephrologist and investigator and who are willing to stop (Parts A and B) or reduce (Part C) their stable ESA dose from the week of randomization until completion of the 6-week treatment period (unless rescue therapy is needed)
* Have a hemoglobin value (taken prior to dialysis if taken on a dialysis day) greater than or equal to 9.5 grams per deciLiter (g/dL) and less than or equal to 12.5 g/dL at screening
* Have a body mass index (BMI) of 18.5 to 45 kilograms per square meter (kg/m^2) inclusive at screening
* Have a transferrin saturation (TSat) greater than or equality to 15 percent and ferritin greater than 40 nanograms per milliliter (ng/mL) at screening

Exclusion Criteria:

* Any cause of anemia other than renal disease
* A history of hyporesponsiveness to ESA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Davita Clinical Research, DN, Lakewood, Colorado
  - Orlando Clinical Research Center, Orlando, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Davita Clinical Research, Minneapolis, Minnesota

REFERENCES:
- [Derived] Sheetz M, Barrington P, Callies S, Berg PH, McColm J, Marbury T, Decker B, Dyas GL, Truhlar SME, Benschop R, Leung D, Berg J, Witcher DR. Targeting the hepcidin-ferroportin pathway in anaemia of chronic kidney disease. Br J Clin Pharmacol. 2019 May;85(5):935-948. doi: 10.1111/bcp.13877. Epub 2019 Mar 4. PMID 30677788

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included three parts. Part A was dose escalation (placebo, 300, 600, or 1,000 milligrams [mg] LY2928057). Part B was dose expansion (placebo or 1000 mg LY2928057). Part C was optional, based on predefined pharmacodynamics criteria. Part C was not executed.
Groups:
- Placebo: Placebo administered intravenously (IV) once every two weeks (Q2W) for six weeks (three doses).
- 300 mg LY2928057: 300 milligrams (mg) LY2928057 administered IV Q2W for six weeks (three doses).
- 600 mg LY2928057: 600 mg LY2928057 administered IV Q2W for six weeks (three doses).
- 1000 mg LY2928057: 1000 mg LY2928057 administered IV Q2W for six weeks (three doses).
Period: Dose Level: Placebo
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Started | 7 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 7 | 0 | 0 | 0
Completed | 7 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Dose Level 300 mg
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Started | 0 (Multiple periods were added for each dose level to represent dose escalation.) | 6 (Multiple periods were added for each dose level to represent dose escalation.) | 0 | 0
Received at Least One Dose of Study Drug | 0 | 6 | 0 | 0
Completed | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Dose Level 600 mg
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Started | 0 | 0 (Multiple periods were added for each dose level to represent dose escalation.) | 11 (Multiple periods were added for each dose level to represent dose escalation.) | 0
Receive at Least One Dose of Study Drug | 0 | 0 | 11 | 0
Completed | 0 | 0 | 9 | 0
Not Completed | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Period: Dose Level 1000 mg
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Started | 0 | 0 | 0 (Multiple periods were added for each dose level to represent dose escalation.) | 4 (Multiple periods were added for each dose level to represent dose escalation.)
Received at Least One Dose of Study Drug | 0 | 0 | 0 | 4
Completed | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Placebo: Placebo administered IV Q2W for six weeks (three doses).
- 300 mg LY2928057: 300 mg LY2928057 administered IV Q2W for six weeks (three doses).
- Total: Total of all reporting groups
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057 | Total
Number analyzed (Participants) | 7 | 6 | 11 | 4 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (9.1) | 52.5 (4.1) | 52.5 (7.6) | 61.0 (9.8) | 53.6 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 2 | 9
  Male | 5 | 4 | 8 | 2 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 0 | 3
  Not Hispanic or Latino | 6 | 6 | 9 | 4 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 7 | 3 | 19
  White | 3 | 1 | 4 | 1 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 11 | 4 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of other nonserious adverse events (AEs) and all SAEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline to Study Completion (up to Day 137)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 7 | 6 | 11 | 4
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Hemoglobin at 6 Week Endpoint
Time Frame: Baseline, Day 42
Population: All participants who received three doses of study drug, had pharmacodynamics assessment at Week 6, and/or received anti-anemic rescue therapy per protocol, regardless of whether they completed treatment.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 7 | 5 | 9 | 2
grams per deciliter (g/dL) | -1.674 (0.5535) | -1.739 (0.5261) | -0.906 (0.4577) | -1.623 (1.0469)

3. Secondary Outcome: Pharmacodynamics (PD): Maximum Change in Hemoglobin
Time Frame: Baseline through 6 Weeks
Population: All participants who received at least one dose of study drug had evaluable hemoglobin values at baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: millimoles per liter of iron (mml/L-Fe)
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 7 | 6 | 11 | 4
millimoles per liter of iron (mml/L-Fe) | 1.294 (0.320) | 1.677 (0.701) | 1.162 (0.367) | 1.348 (0.563)

4. Secondary Outcome: Pharmacodynamics (PD): Geometric Mean Ratio of Serum Iron (Fe) Concentrations Relative to Baseline
Description: Pharmacodynamics (PD): Geometric Mean Ratio of Serum Iron (Fe) Concentrations relative to baseline.
Time Frame: Baseline, 6 weeks
Population: All participants who received at least one dose of study drug and had evaluable serum Fe values at baseline and post-baseline.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 7 | 6 | 11 | 4
Ratio | 0.99 (16) | 1.57 (32) | 1.59 (69) | 2.36 (44)

5. Secondary Outcome: Pharmacodynamics (PD): Maximum Change in Transferrin Saturation (TSat)
Time Frame: Baseline through 6 weeks
Population: All participants who received at least one dose of study drug and had evaluable TSat values at baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: percentage change in TSat
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 6 | 6 | 9 | 4
percentage change in TSat | 0.2117 (0.1120) | 0.5250 (0.0873) | 0.5000 (0.1550) | 0.4375 (0.0624)

6. Secondary Outcome: Pharmacodynamics (PD): Maximum Change in Concentration of Hemoglobin in Reticulocytes (CHr)
Time Frame: Baseline through 6 weeks
Population: All participants who received at least one dose of study drug had evaluable CHr values at baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: picograms (pg)
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 7 | 6 | 11 | 4
picograms (pg) | 1.93 (0.45) | 3.00 (1.18) | 3.60 (2.31) | 3.20 (1.45)

7. Secondary Outcome: Pharmacodynamics (PD): Maximum Change in Reticulocyte Count
Time Frame: Baseline through 6 weeks
Population: All participants who received at least one dose of study drug and had evaluable reticulocyte values at baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: gigaparticles per liter (GI/L)
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 7 | 6 | 11 | 2
gigaparticles per liter (GI/L) | 49 (37.6) | 72.17 (29.21) | 40.73 (13.81) | 74.25 (78.73)

8. Secondary Outcome: Pharmacodynamics (PD): Maximum Change in Red Blood Cell (RBC) Count
Time Frame: Baseline through 6 weeks
Population: All participants who received at least one dose of study drug and had evaluable RBC values at baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: tera per liter (TI/L)
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 7 | 6 | 11 | 4
tera per liter (TI/L) | 0.686 (0.135) | 0.900 (0.341) | 0.627 (0.228) | 0.725 (0.299)

9. Secondary Outcome: Pharmacodynamics (PD): Maximum Change in Mean Corpuscular Volume (MCV)
Time Frame: Baseline through 6 weeks
Population: All participants who received at least one dose of study drug and had evaluable MCV values at baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: femtoliters (fL)
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 7 | 6 | 11 | 4
femtoliters (fL) | 5.9 (4.6) | 5.2 (1.9) | 6.2 (1.7) | 7.0 (3.2)

10. Secondary Outcome: Pharmacodynamics (PD): Maximum Change in Mean Corpuscular Hemoglobin (MCH)
Time Frame: Baseline through 6 weeks
Population: All participants who received at least one dose of study drug and had evaluable MCH values at baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: femtomoles of iron (fmol[Fe])
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 7 | 6 | 11 | 4
femtomoles of iron (fmol[Fe]) | 0.107 (0.029) | 0.105 (0.027) | 0.091 (0.050) | 0.080 (0.034)

11. Secondary Outcome: Pharmacodynamics (PD): Maximum Change in Mean Corpuscular Hemoglobin Concentration (MCHC)
Time Frame: Baseline through 6 weeks
Population: All participants who received at least one dose of study drug and had evaluable MCHC values at baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: millimoles/liter of iron (mml/L-Fe)
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 7 | 6 | 11 | 4
millimoles/liter of iron (mml/L-Fe) | 1.4 (0.5) | 1.2 (0.4) | 1.6 (0.7) | 1.5 (0.6)

12. Secondary Outcome: Pharmacodynamics (PD): Maximum Change in Ferritin
Time Frame: Baseline through 6 weeks
Population: All participants who received at least one dose of study drug and had evaluable ferritin values at baseline and post-baseline.
Measure: Mean (Standard Deviation); unit: micrograms/liter (ug/L)
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 7 | 6 | 11 | 4
micrograms/liter (ug/L) | 269.21 (112.17) | 230.28 (80.08) | 196.46 (90.90) | 146.65 (48.05)

13. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2928057
Description: Time frame for Cycle 2: Predose, end of infusion, prior to end of dialysis or 2h, post dialysis or 4h, 2 days (d), 4d, 7d, 9d, 11d postdose;
  Time frame for Cycle 3: Predose, end of infusion, prior to end of dialysis or 2h, post dialysis or 4h, 2d, 4d, 7d, 9d, 11d, 14d postdose
Time Frame: Cycle 1: Predose, end of infusion, 2hours(h), 4h, 2d, 4d, 7d, 9d, 11d postdose;
Population: All participants who received at least one dose of LY2928057 and had evaluable plasma values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 6 | 11 | 4
micrograms per milliliter (µg/mL)
  Cycle 1 (First dose) | 67.3 (25) | 274 (104) | 312 (21)
  Cycle 2 (Second dose) | 70.0 (21) | 213 (49) | 397 (30)
  Cycle 3 (Third dose): number analyzed (Participants) | 6 | 8 | 2
  Cycle 3 (Third dose) | 62.8 (21) | 177 (34) | 358 (NA) — Coefficient of variation was not produced as there are only 2 participants.

14. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve From Time Zero to Infinity (AUC[0-inf]) of LY2928057
Description: Time frame for Cycle 2: Predose, end of infusion, prior to end of dialysis or 2h, post dialysis or 4h, 2d, 4d, 7d, 9d, 11d postdose;
  Time frame for Cycle 3: Predose, end of infusion, prior to end of dialysis or 2h, post dialysis or 4h, 2d, 4d, 7d, 9d, 11d, 14d postdose;
Time Frame: Cycle 1: Predose, end of infusion, 2hours(h), 4h, 2d, 4d, 7d, 9d, 11d postdose
Population: All participants who received at least one dose of LY2928057 and had evaluable plasma values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms x hours/milliliter(µg*h/mL)
Arm/Group | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 6 | 11 | 4
micrograms x hours/milliliter(µg*h/mL)
  Cycle 1 (First dose) | 1560 (39) | 7340 (33) | 11200 (24)
  Cycle 2 (Second dose) | 1640 (42) | 6970 (40) | 16100 (31)
  Cycle 3 (Third dose): number analyzed (Participants) | 6 | 8 | 2
  Cycle 3 (Third dose) | 1520 (40) | 6520 (25) | 12000 (NA) — Coefficient of variation was not produced as there are only 2 participants.

15. Secondary Outcome: Number of Participants With Anti-LY2928057 Antibodies
Time Frame: Baseline through 84 days
Population: All participants who received at least one dose of study drug and had evaluable antibody values at baseline and post-baseline.
Measure: Number; unit: participants
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 7 | 6 | 11 | 4
participants | 1 | 4 | 6 | 3

16. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From 0 to 336 Hours AUC(0-336) During and Outside Dialysis
Description: Time frame for Cycle 2: Predose, end of infusion, prior to end of dialysis or 2h, post dialysis or 4h, 2d, 4d, 7d, 9d, 11d postdose;
  Dialysis did not occur in cycle 1.
Time Frame: Cycle 1: Predose, end of infusion, 2hours, 4h, 2d, 4d, 7d, 9d, 11d postdose
Population: All participants who received 300 mg LY2928057 or 600 mg LY2928057 during dialysis and non-dialysis day and had evaluable plasma values. Data were not collected in the 1000 mg LY2928057 arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | 300 mg LY2928057 | 600 mg LY2928057
Number analyzed (Participants) | 6 | 11
hr*ng/mL
  Cycle 1 (First dose, no dialysis) | 1550 (39) | 7320 (33)
  Cycle 2 (Second dose during dialysis) | 1630 (42) | 6940 (40)

ADVERSE EVENTS:
Arm/Group | Placebo | 300 mg LY2928057 | 600 mg LY2928057 | 1000 mg LY2928057
Serious Adverse Events (participants affected / at risk) | 0/7 | 2/6 | 0/11 | 1/4
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 8/11 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | 300 mg LY2928057 (N=6) | 600 mg LY2928057 (N=11) | 1000 mg LY2928057 (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | 300 mg LY2928057 (N=6) | 600 mg LY2928057 (N=11) | 1000 mg LY2928057 (N=4)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 2 (2) | 3 (3) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days